CLINICAL TRIAL: NCT03280394
Title: Prospective, Observational, Multi-centred, Non-interventional Research Project on Plasma Cell Free DNA Genotyping as a Tool to Inform Mature B-cell Tumor Management
Brief Title: Liquid Biopsy in Mature B-cell Tumors
Status: Recruiting | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Davide Rossi, MD, PhD, Oncology Institute of Southern Switzerland
Other Study IDs: IOSI-EMA003
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Mature B-Cell Neoplasm
Keywords: Liquid biopsy; Classical Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Mutations
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell | interventions — Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (20 ml in EDTA tubes and 20 ml in Cell-Free DNA BCT tubes)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Liquid Biopsy — Assessing whether plasma cell free DNA improves the accuracy of early prediction of cure in mature B-cell tumor patients and whether it represents an accessible source of tumor DNA for the sensitive identification of genetic biomarkers that, at disease presentation, refine the diagnostic workup in mature B-cell tumor patients and, upon treatment, early identify the emergence of resistance mutations.

SUMMARY:
The study aims at assessing whether cell free DNA genotyping can improve the accuracy of early prediction of cure in mature B-cell tumor patients and whether it represents an accessible source of tumor DNA for the sensitive identification of genetic biomarkers that refine the diagnostic workup, stratify prognosis and identify the emergence of drug-resistance mutations during treatment.

DETAILED DESCRIPTION:
Clinical data and peripheral blood samples (20 ml in EDTA tubes and 20 ml in Cell-Free DNA BCT tubes) will be collected during the clinico/laboratory visits that are planned as per clinical routine at the time of mature B-cell tumor diagnosis, before treatment, at the time of interim PET/CT, at the time of end of treatment PET/CT and at the time of disease relapse.

Clinical variables, international prognostic index, results of plasma cell free DNA genotyping and of PET-CT will be analyzed descriptively.

The sensitivity, specificity, positive predictive value, negative predictive value and accuracy of the compiled results of plasma cell free DNA genotyping and interim PET-CT (for cHL and DLBCL), or plasma cell free DNA genotyping and baseline international prognostic index (for FL and MCL) in identifying patients that are progression free for >24 months after first line therapy will be calculated and compared with those obtained by the sole interim PET-CT (cHL and DLBCL) or the sole international prognostic index (FL, MCL).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 years or older
* Documented diagnosis of mature B-cell tumor according to WHO 2008 criteria
* Willing and able to comply with scheduled study procedures
* Evidence of a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female adults 18 years or older with a documented diagnosis of mature B-cell tumor according to WHO 2008 criteria
Sampling Method: Non-Probability Sample
Enrollment: 444 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of interim plasma cell free DNA genotyping for cHL patients | 24 months from treatment
  Assessment of interim plasma cell free DNA genotyping accuracy in the identification of cured vs non cured patients in cHL (patients not progressed after 24 months)
Accuracy of interim plasma cell free DNA genotyping for DLBCL patients | 24 months from treatment
  Assessment of interim plasma cell free DNA genotyping accuracy in the identification of cured vs non cured patients in DLBCL (patients not progressed after 24 months)
Accuracy of interim plasma cell free DNA genotyping for FL patients | 24 months from treatment
  Assessment of interim plasma cell free DNA genotyping accuracy in the identification of patients in continuous complete remission at 24 months from first line treatment vs patients not in continuous complete remission at 24 months from first line treatment in FL and other indolent B-cell lymphoproliferative disorders
Accuracy of interim plasma cell free DNA genotyping for MCL patients | 24 months from treatment
  Assessment of interim plasma cell free DNA genotyping accuracy in the identification of patients in continuous complete remission at 24 months from first line treatment vs patients not in continuous complete remission at 24 months from first line treatment in MCL

CONTACTS AND LOCATIONS:
Overall Officials: Davide Rossi, MD, PhD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (1):
- Institute of Oncology Research, Bellinzona, Canton Ticino, Switzerland